CLINICAL TRIAL: NCT03016624
Title: Coronary Artery Healing Process After BiOresorbable Scaffold iN PatiEnts With Non-ST-Segment Elevation Myocardial Infarction (NSTEMI)
Brief Title: Coronary Artery Healing and Bioresorbable Scaffold
Acronym: HONEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Christian Oliver Fallesen, MD, PhD student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20150133
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCT guided Magmaris implantation (Active Comparator): Percutaneous coronary intervention with Magmaris
  Interventions: Device: OCT guided PCI
- Angiography guided Magmaris implantation (Active Comparator): Percutaneous coronary intervention with Magmaris
  Interventions: Device: Angiography guided PCI

INTERVENTIONS:
Device: OCT guided PCI — oct guided
  Arms: OCT guided Magmaris implantation
Device: Angiography guided PCI — angio guided
  Arms: Angiography guided Magmaris implantation

SUMMARY:
To compare coronary healing after optical coherence tomography guided versus conventionally angiography guided percutaneous coronary intervention with the Magmaris bioresorbable scaffold.

DETAILED DESCRIPTION:
BACKGROUND:

Bioresorbable scaffolds (BRS) represent a novel approach during percutaneous coronary intervention (PCI), which provides transient vessel support with drug-delivery capability without the long-term limitations (very late stent thrombosis) of the metallic drug-eluting stents. Patients with Non-ST-segment elevation myocardial infarction (NSTEMI) often feature thrombus-rich lesions with large necrotic core, which may be associated with delayed arterial healing and impaired stent-related outcomes. Besides clinical indication and underlying plaque morphology, sufficient and potent strut coverage depends on several additional factors (patient characteristics, stent type and procedural factors). Particularly, acute incomplete stent apposition is a strong procedural risk factor for later deficient neointimal coverage. Optical coherence tomography (OCT) is a high-resolution intravascular imaging modality, that enables in-vivo evaluation of the immediate stenting result, and the vascular healing pattern including strut coverage at follow-up.

AIM:

The objective of this study is to investigate if OCT-guided Magmaris BRS implantation in patients with NSTEMI can improve the coronary arterial healing at 6 months compared to routine angiographic guidance only. Further to investigate if the plaque composition/lipid content will influence on the vascular healing.

METHOD:

The study is designed as a prospective, randomized trial. After pre-dilation, patients will be randomly assigned to either: (1) OCT-guided PCI, or (2) angio-guided PCI with Magmaris BRS implantation. In the OCT-guided group, OCT will be used for vessel and BRS sizing. After Magmaris BRS implantation the result will be controlled with OCT and: 1) BRS under expansion and/or, 2) strut malapposition and/or, 3) edge dissection- and/or 4) residual stenosis at the distal and/or proximal reference segment(s) that may require further intervention. A final OCT will be performed in case of re-intervention.

In the angio-guided group an OCT will be performed only after angiography final and acceptable result.

A follow-up OCT will be performed after 6 months in all patients to assess the vascular healing and a vasomotor test will be performed in half of the patients. After 12 months the dynamic changes in vascular healing will be assessed in the first enrolled half of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSTEMI undergoing subacute PCI in native vessels and to be treated with one or more drug eluting stents in coronary arteries due to a visually assessed significant culprit lesion with > 50% of coronary stenosis at the catheterization laboratory in Odense.

Exclusion Criteria:

* Patients participating in other randomized stent studies.
* Expected survival < 1 year.
* Allergy to aspirin, ticagrelor, clopidogrel and prasugrel.
* Allergy to Sirolimus.
* Aorta-ostial lesions (cannot be cleared with flush by OCT).
* Serum creatinine > 150 ug/L due to the required amount of X-ray contrast by OCT.
* Twisted coronary vessels where the PCI-operator estimates that the introduction of an OCT and / or NIRS catheter will not be possible or will be associated with increased risk.
* Lesion length > 28 mm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Coronary artery healing score | 6 months
  The primary endpoint is coronary artery healing score assessed by OCT Healing score is a weighted index that combines the following components: Uncovered scaffold struts, Uncovered "jailed" and acquired or persistent malapposed struts, Persistent mal apposition, Acquired mal apposition, Maximum neointimal growth and Accumulated extra stent lumen

SECONDARY OUTCOMES:
Coronary artery healing | 6 and 12 months.
  Secondary endpoints are all individual components of coronary artery healing score
Coronary artery healing | 6 months
  Vasomotion at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisette O Jensen, MD, DMSci, PhD, Professor, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark

REFERENCES:
- [Derived] Fallesen CO, Antonsen L, Maehara A, Noori M, Hougaard M, Hansen KN, Ellert J, Ahlehoff O, Veien KT, Lassen JF, Junker AB, Hansen HS, Jensen LO. Optical Coherence Tomography- Versus Angiography-Guided Magnesium Bioresorbable Scaffold Implantation in NSTEMI Patients. Cardiovasc Revasc Med. 2022 Jul;40:101-110. doi: 10.1016/j.carrev.2021.12.003. Epub 2021 Dec 15. PMID 34949544